CLINICAL TRIAL: NCT05382351
Title: Exploratory Study on Antiviral Therapy for Patients With Chronic Hepatitis B Virus Infection (Immune Tolerance Period)
Brief Title: Antiviral Therapy for Patients With Chronic Hepatitis B Infection
Status: Unknown | Phase: Phase 2 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Sun Yat-sen University (Other)
Responsible Party: Principal Investigator, Lin Bingliang, Exploratory study on antiviral therapy for patients with chronic hepatitis B virus infection (immune tolerance period), Sun Yat-sen University
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: Treatment for CHB infection
Record Dates: First submitted 2022-05-15; First posted 2022-05-19 (Actual); Last update posted 2022-05-19 (Actual); Status verified 2022-05

CONDITIONS: Chronic Hepatitis B Virus Infection
MeSH Terms: conditions — Hepatitis B, Chronic | interventions — entecavir

STUDY DESIGN:
Who Masked: Investigator
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Entecavir group (Experimental): Patients receive treatment with entecavir
  Interventions: Drug: Entecavir
- Entecavir and Tenofovir Amibufenamide group (Experimental): Patients will receive the treatment of entecavir combined with tenofovir amibufenamide
  Interventions: Drug: Entecavir combined with Tenofovir Amibufenamide

INTERVENTIONS:
Drug: Entecavir — Entecavir group will receive entecavir orally once a day, 0.5mg each time, and fasting for 2h before and after taking the medicine
  Other Names: Boludine/Rui fu en
  Arms: Entecavir group
Drug: Entecavir combined with Tenofovir Amibufenamide — Entecavir combined with Tenofovir Amibufenamide group will be treated with entecavir and tenofovir amibufenamide. Entecavir is administered in the same way as before. enofovir amibufenamide orally 25mg once a day with meals
  Other Names: Heng mu
  Arms: Entecavir and Tenofovir Amibufenamide group

SUMMARY:
The study aims to demonstrate that antiviral therapy for patients with immune tolerance of CHB. On the basis of the original antiviral therapy of entecavir, further clarify the safety and effectiveness of entecavir combined with tenofovir amibufenamide.The investigators plan to enroll about 328 hepatitis B patients,. who are in the stage of immune tolerance. These participants will be devided into two groups randomly .Group A will receive the treatment of entecavir. Group B will be treated with entecavir and tenofovir amibufenamide. The participants in both groups will be followed up for 96 weeks.

The primary endpoint is to compare the inhibition rate of HBV-DNA between two groups. The secondary endpoint includes: (1) Comparing the decrease of HBV DNA at 48 weeks between the two groups. (2) Comparing the HBeAg seroconversion rates at 48 weeks and 96 weeks between the two groups. (3) The changes of HBsAg at 48 weeks and 96 weeks between the two groups. (4) Comparing adverse side effects between the two groups.

DETAILED DESCRIPTION:
High HBV DNA level is an independent risk factor for liver cirrhosis and liver cancer, we know all patients with chronic hepatitis B virus infection in immune tolerance period had high viral load. So it is necessary to implement antiviral therapy for patients with chronic hepatitis B virus infection in immune tolerance period.Previous studies have found that combination of two antiviral drugs has a higher virological inhibition rate in patients with high viral load than single drug. Hence, the investigators' hypothesis is that treatment of patients with chronic hepatitis B virus infection in immune tolerance period result in higher virological inhibition rate and reduce of the risk of cirrhosis and liver cancer.

The investigators plan to enroll about 328 hepatitis B patients, who are in the stage of immune tolerance. These participants will be devided into 2 groups.Group A will receive the treatment of entecavir . Group B will be treated with entecavir and tenofovir amibufenamide. The participants in both groups will be followed up for 96 weeks. Unless there are serious adverse drug reactions, the protocol cannot be adjusted within 96 weeks.

The primary endpoint is to compare the inhibition rate of HBV-DNA between two groups. The secondary endpoint includes: (1) Comparing the decrease of HBV DNA at 48 weeks between the two groups. (2) Comparing the HBeAg seroconversion rates at 48 weeks and 96 weeks between the two groups. (3) The changes of HBsAg at 48 weeks and 96 weeks between the two groups. (4) Comparing adverse side effects between the two groups.

ELIGIBILITY:
Inclusion Criteria:

1. Age between 18-65 years old;
2. HBsAg positive >6 months, HBsAg>1*10e4IU/ml;
3. HBV-DNA> 2 * 10e7IU / ml;
4. HBeAg positive;
5. ALT / AST remained normal which were followed up twice within 1 year with at least a 6-month interval each time.
6. No antiviral treatment with interferon or nucleoside (acid) analogues in the previous year

Exclusion Criteria:

1. infection with hepatitis A, C, D, E viruses or HIV infection ;
2. Combined with diabetes, hypertension, renal insufficiency, autoimmune diseases and other organ dysfunction And malignant tumors;
3. Patients using Immunosuppressive therapy or radiotherapy / chemotherapy for other diseases;
4. Patients with liver fibrosis, cirrhosis (FibroScan > = 9.4kpa) and liver cancer were identified;
5. Extrahepatic manifestations related to HBV (glomerulonephritis, vasculitis, nodular polyarteritis, peripheral neuropathy, etc.);
6. Allergic to nucleoside drugs
7. Pregnancy or having pregnancy plan within 2 years and Lactating patients;
8. Patients who are unable to comply with the arrange ment of this study or sign the informed consent.
9. Failed to return to hospital regularly for follow-up ac- cording to the study plan.
10. Researchers determine other condition that does not fit into the study.

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 238 (Estimated)
Dates: Start 2022-05-10 (Actual); Primary Completion 2024-04-30 (Estimated); Study Completion 2024-12-31 (Estimated)

PRIMARY OUTCOMES:
The inhibition rate of HBV-DNA between two groups | 96 weeks
  compare the inhibition rate of HBV-DNA between two groups at 96 weeks

SECONDARY OUTCOMES:
The decrease of HBV DNA in the at 48 weeks between the two groups | 48 weeks
  comparing the decrease of HBV DNA in the at 48 weeks between the two groups
The HBeAg seroconversion rates at 48 weeks and 96 weeks | 48 weeks and 96 weeks
  comparing the HBeAg seroconversion rates at 48 weeks and 96 weeks between the two groups
The changes of HBsAg | 48 weeks and 96 weeks
  The changes of HBsAg at 48 weeks and 96 weeks were compared between the two groups
adverse side effects | 4、12、24、48、72 and 96 weeks
  comparing adverse side effects between the two groups

CONTACTS AND LOCATIONS:
Locations (1):
- The Third Affiliated Hospital of Sun Yat-sen University, Guangzhou, Guangdong, China

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Fattovich G, Bortolotti F, Donato F. Natural history of chronic hepatitis B: special emphasis on disease progression and prognostic factors. J Hepatol. 2008 Feb;48(2):335-52. doi: 10.1016/j.jhep.2007.11.011. Epub 2007 Dec 4. PMID 18096267
- [Background] Lok AS, McMahon BJ. Chronic hepatitis B. Hepatology. 2007 Feb;45(2):507-39. doi: 10.1002/hep.21513. No abstract available. PMID 17256718
- [Background] Chen CJ, Yang HI, Su J, Jen CL, You SL, Lu SN, Huang GT, Iloeje UH; REVEAL-HBV Study Group. Risk of hepatocellular carcinoma across a biological gradient of serum hepatitis B virus DNA level. JAMA. 2006 Jan 4;295(1):65-73. doi: 10.1001/jama.295.1.65. PMID 16391218
- [Background] Tang LSY, Covert E, Wilson E, Kottilil S. Chronic Hepatitis B Infection: A Review. JAMA. 2018 May 1;319(17):1802-1813. doi: 10.1001/jama.2018.3795. PMID 29715359
- [Background] Raffetti E, Fattovich G, Donato F. Incidence of hepatocellular carcinoma in untreated subjects with chronic hepatitis B: a systematic review and meta-analysis. Liver Int. 2016 Sep;36(9):1239-51. doi: 10.1111/liv.13142. Epub 2016 May 22. PMID 27062182
- [Background] Chayanupatkul M, Omino R, Mittal S, Kramer JR, Richardson P, Thrift AP, El-Serag HB, Kanwal F. Hepatocellular carcinoma in the absence of cirrhosis in patients with chronic hepatitis B virus infection. J Hepatol. 2017 Feb;66(2):355-362. doi: 10.1016/j.jhep.2016.09.013. Epub 2016 Sep 28. PMID 27693539
- [Background] Wong GL, Chan HL, Chan HY, Tse PC, Tse YK, Mak CW, Lee SK, Ip ZM, Lam AT, Iu HW, Leung JM, Wong VW. Accuracy of risk scores for patients with chronic hepatitis B receiving entecavir treatment. Gastroenterology. 2013 May;144(5):933-44. doi: 10.1053/j.gastro.2013.02.002. Epub 2013 Feb 12. PMID 23415803
- [Background] Kumar M, Sarin SK, Hissar S, Pande C, Sakhuja P, Sharma BC, Chauhan R, Bose S. Virologic and histologic features of chronic hepatitis B virus-infected asymptomatic patients with persistently normal ALT. Gastroenterology. 2008 May;134(5):1376-84. doi: 10.1053/j.gastro.2008.02.075. Epub 2008 Feb 29. PMID 18471514
- [Background] Wong GL, Wong VW, Choi PC, Chan AW, Chim AM, Yiu KK, Chan HY, Chan FK, Sung JJ, Chan HL. Clinical factors associated with liver stiffness in hepatitis B e antigen-positive chronic hepatitis B patients. Clin Gastroenterol Hepatol. 2009 Feb;7(2):227-33. doi: 10.1016/j.cgh.2008.10.023. Epub 2008 Oct 30. PMID 19121647
- [Background] Seto WK, Lai CL, Ip PP, Fung J, Wong DK, Yuen JC, Hung IF, Yuen MF. A large population histology study showing the lack of association between ALT elevation and significant fibrosis in chronic hepatitis B. PLoS One. 2012;7(2):e32622. doi: 10.1371/journal.pone.0032622. Epub 2012 Feb 28. PMID 22389715
- [Background] Lok AS, McMahon BJ, Brown RS Jr, Wong JB, Ahmed AT, Farah W, Almasri J, Alahdab F, Benkhadra K, Mouchli MA, Singh S, Mohamed EA, Abu Dabrh AM, Prokop LJ, Wang Z, Murad MH, Mohammed K. Antiviral therapy for chronic hepatitis B viral infection in adults: A systematic review and meta-analysis. Hepatology. 2016 Jan;63(1):284-306. doi: 10.1002/hep.28280. Epub 2015 Nov 13. PMID 26566246
- [Background] Wong GL, Wong VW, Chan HY, Tse PC, Wong J, Chim AM, Yiu KK, Chu SH, Chan HL. Undetectable HBV DNA at month 12 of entecavir treatment predicts maintained viral suppression and HBeAg-seroconversion in chronic hepatitis B patients at 3 years. Aliment Pharmacol Ther. 2012 Jun;35(11):1326-35. doi: 10.1111/j.1365-2036.2012.05098.x. Epub 2012 Apr 16. PMID 22506552
- [Background] Wong GL, Chan HL, Mak CW, Lee SK, Ip ZM, Lam AT, Iu HW, Leung JM, Lai JW, Lo AO, Chan HY, Wong VW. Entecavir treatment reduces hepatic events and deaths in chronic hepatitis B patients with liver cirrhosis. Hepatology. 2013 Nov;58(5):1537-47. doi: 10.1002/hep.26301. Epub 2013 Sep 30. PMID 23389810
- [Background] Zoutendijk R, Reijnders JG, Zoulim F, Brown A, Mutimer DJ, Deterding K, Hofmann WP, Petersen J, Fasano M, Buti M, Berg T, Hansen BE, Sonneveld MJ, Wedemeyer H, Janssen HL; VIRGIL Surveillance Study Group. Virological response to entecavir is associated with a better clinical outcome in chronic hepatitis B patients with cirrhosis. Gut. 2013 May;62(5):760-5. doi: 10.1136/gutjnl-2012-302024. Epub 2012 Apr 5. PMID 22490523
- [Background] Lok AS, Trinh H, Carosi G, Akarca US, Gadano A, Habersetzer F, Sievert W, Wong D, Lovegren M, Cohen D, Llamoso C. Efficacy of entecavir with or without tenofovir disoproxil fumarate for nucleos(t)ide-naive patients with chronic hepatitis B. Gastroenterology. 2012 Sep;143(3):619-628.e1. doi: 10.1053/j.gastro.2012.05.037. Epub 2012 May 27. PMID 22643350
- [Background] Chan HL, Chan CK, Hui AJ, Chan S, Poordad F, Chang TT, Mathurin P, Flaherty JF, Lin L, Corsa A, Gaggar A, Subramanian GM, McHutchison JG, Lau G, Lee S, Gane EJ. Effects of tenofovir disoproxil fumarate in hepatitis B e antigen-positive patients with normal levels of alanine aminotransferase and high levels of hepatitis B virus DNA. Gastroenterology. 2014 May;146(5):1240-8. doi: 10.1053/j.gastro.2014.01.044. Epub 2014 Jan 23. PMID 24462735
- [Background] Mauss S, Berger F, Filmann N, Hueppe D, Henke J, Hegener P, Athmann C, Schmutz G, Herrmann E. Effect of HBV polymerase inhibitors on renal function in patients with chronic hepatitis B. J Hepatol. 2011 Dec;55(6):1235-40. doi: 10.1016/j.jhep.2011.03.030. Epub 2011 May 19. PMID 21703180
- [Background] Duarte-Rojo A, Heathcote EJ. Efficacy and safety of tenofovir disoproxil fumarate in patients with chronic hepatitis B. Therap Adv Gastroenterol. 2010 Mar;3(2):107-19. doi: 10.1177/1756283X09354562. PMID 21180595